CLINICAL TRIAL: NCT04855799
Title: Direct Measurement of Gastrointestinal Permeability Change in Response to Aquamin®
Brief Title: GI Permeability Change in Response to Aquamin®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James Varani (Other)
Responsible Party: Sponsor-Investigator, James Varani, Professor of Pathology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00156676 sub-study 1
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis; Healthy; Irritable Bowel Syndrome With Diarrhea
Keywords: gastrointestinal permeability
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Aquamin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aquamin® (Experimental)
  Interventions: Drug: Aquamin

INTERVENTIONS:
Drug: Aquamin — Participants will take a 90-day supply of Aquamin®, 4 capsules per day; 2 to be taken in the morning and 2 in the evening (containing approximately 800 mg calcium/day).
  Other Names: Nutritional

SUMMARY:
This trial is being completed to learn about how Aquamin® affects gastrointestinal permeability, or the control of material passing from inside the gastrointestinal tract through the gut wall into the rest of the body, in people with ulcerative colitis (UC), Irritable Bowel Syndrome with diarrhea (IBS-D), and in healthy individuals.

DETAILED DESCRIPTION:
This is a sub-study to the ongoing clinical trial entitled: Aquamin®, a multi-mineral natural product from red marine algae, as an adjuvant intervention for mild ulcerative colitis and ulcerative colitis in remission (HUM00156676) NCT# NCT03869905.

ELIGIBILITY:
Inclusion Criteria for UC participants:

* Must be able to give written informed consent
* Age 18 to 80 years old.
* Must have: Ulcerative colitis with confirmed diagnosis by histology and endoscopy; and be in stable remission for 3 months or more without therapy or with maintenance therapy (except steroids and antibiotics for 3 months) or have mild ulcerative colitis. Note: Corticosteroids (a type of steroid drug such as prednisone or cortisol that helps the body to regulate stress response, immune response and inflammation) and antibiotics can be used during a flare-up once the study has begun and the subject enrolled.
* A negative pregnancy test for pre-menopausal women with intact female reproductive organs. Must agree to use appropriate birth control over the study period (if applicable).

If cessation of menses is within 12 months, then the participant will be treated as pre-menopausal and a pregnancy test will be performed.

Inclusion Criteria for Healthy participants:

* Must be able to give written informed consent
* Be generally healthy, male or female, ages 18 to 80 years old.
* Pre-menopausal women with intact female reproductive organs must have a negative pregnancy test within 2 weeks of the Baseline Visit.
* Subject must agree to use appropriate birth control over the study period. (Post-menopausal is defined as no menses for the previous 12 months. If cessation of menses is within 12 months, then the participant will be treated as pre-menopausal and a pregnancy test will be performed.

Inclusion Criteria for participants with IBS-D:

* Patients with ages 18-80 years old.
* Must meet the IBS-D Diagnostic Rome IV (four) Criteria as noted in the protocol
* A negative pregnancy test for pre-menopausal cis-women with intact vagina, uterus, and/or ovaries. The negative pregnancy test must be within 2 weeks of the baseline visit and the subject must agree to use appropriate birth control over the study period.

Exclusion Criteria For UC participants:

* Must not be pregnant or lactating
* Must not be participating in any other interventional trial using an investigational drug.
* Subjects likely to be uncooperative or unable to comply with study procedures
* Participants must not be felt to have active ulcerative colitis for 3 months before study enrollment (with an exception of mild ulcerative colitis).
* Participants must not have a history or diagnosis of any of the following conditions:

Crohn's disease, Any stomach or intestinal bleeding disorders (gastrointestinal bleeding from gastric or duodenal ulcers, or gastrin secreting tumors) or active gastric/duodenal ulcers - peptic ulcer disease (without bleeding in last 3 months).

* Must not have any gastrointestinal or colonic malignancy.
* Must not have Kidney disease, including kidney "stones" or hypercalcemia.
* Must not have Coagulopathy/hereditary hemorrhagic disorders
* Participants will be excluded if they have taken certain medications (per protocol), within the last 30 days or are unwilling to forgo the following for 30 days prior to entry into the study.

Exclusion Criteria For Healthy participants:

* Must not be pregnant or lactating.
* Must not be participating in any other interventional trial using an investigational drug.
* Participants must not have a history or diagnosis of any of the following conditions:

Kidney disease, including kidney "stones" or hypercalcemia, Crohn's disease, Neurologic disease, other inflammatory bowel disease, any stomach or intestinal bleeding disorders (gastrointestinal bleeding from gastric or duodenal ulcers, or gastrin secreting tumors) or active gastric/duodenal ulcers - peptic ulcer disease (without bleeding in last 3 months).

* Not have Coagulopathy/hereditary hemorrhagic disorders
* Any gastrointestinal or colonic malignancy.
* Participants will be excluded if they have taken certain medications (per protocol), within the last 30 days or are unwilling to forgo the following for 30 days prior to entry into the study.

Exclusion Criteria for participants with IBS-D:

* Must not be pregnant or lactating
* Must not be participating in any other interventional trial using an investigational drug.
* Participants must not have a history or diagnosis of Crohn's disease or Inflammatory bowel disease, any stomach or intestinal bleeding disorders (gastrointestinal bleeding from gastric or duodenal ulcers, or gastrin secreting tumors) or active gastric / duodenal ulcers - peptic ulcer disease (without bleeding in last 3 months).
* Must not have any gastrointestinal or colonic malignancy.
* Must not have kidney disease, including kidney "stones" or hypercalcemia, Coagulopathy/hereditary hemorrhagic disorders, neurologic disease
* Participants will be excluded if they have taken certain medications (per protocol), within the last 30 days or are unwilling to forgo the following for 30 days prior to entry into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Change in the lactulose:mannitol ratio in urine by comparing values at 90-days (post-intervention) to baseline (pre-intervention) levels. | Baseline (pre-intervention), 90 days (post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: James Varani, Principal Investigator — University of Michigan; Muhammad N Aslam, Study Director — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No